CLINICAL TRIAL: NCT05250258
Title: Telephone Peer Support for New Fathers to Prevent Depressive Symptoms After the Child's Birth
Brief Title: Telephone Peer Support to Prevent Depression Among Fathers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ewa Andersson, adjunct professor, Karolinska Institutet
Other Study IDs: 12016/217 -32
Record Dates: First submitted 2020-11-26; First posted 2022-02-22 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Fathers; Depression
Keywords: Telephone peer support; Depression; Fathers
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- telephone peer support: Telephone peer support from experinenced father to father
  Interventions: Other: Telephone peer support by telephone
- Routine care: Standard care as usual in child health care, one visit for fathers and nothing added

INTERVENTIONS:
Other: Telephone peer support by telephone — Peer support by telephone from experienced father to new father with depressive symtoms.
  4 times or more if requested during 4 months
  Groups: telephone peer support

SUMMARY:
The overall purpose of the pilot study is to investigate whether telephone support from fathers to fathers reduces depressive symptoms and stress among new fathers in Sweden. Forty expectant fathers with the Edinburgh Postnatal Depression Scale (EPDS)> 10 two weeks after the birth of the child are divided into two groups where half are allocated to telephone support by other fathers (intervention) as a complement to existing parental support, other group get traditionally existing parental support (control). The fathers in the intervention group were allocated telephone-based support from volunteers who have father experience, not mental illness and have undergone training through this project. These volunteers will be trained and supported by trained mentors. Four months after the child is born, data is collected with questionnaires. The intervention group will be compared with the control group and the results from the pilot study form the basis for the forthcoming RCT. Karolinska Institutet's ethics committee has approved the study. Clinical relevance: The long-term goal of this project is to improve the methods for reducing mental illness among fathers, which leads to a positive development for their children and can be used in the development of clinical guidelines to identify and reduce fathers' stress and depressive symptoms.

DETAILED DESCRIPTION:
The overall aim of the present study is to examine if telephone based peer support to fathers can reduce or prevent depressive symptoms among new fathers in Sweden. Primary outcome: Depressive symptoms, measured by EPDS (Edinburg Postnatal Depression Scale).

Study hypothesis:

It is hypothesized that the provision of telephone-based peer support will reduce depressive symptoms and anxiety among fathers.

Design and methods A pilot controlled clinical trial will be conducted and the different steps are built upon earlier developed peer support.

Fathers will be assigned to telephone based peer support by a coordinator. In this study, fathers will be linked with a peer volunteer during the first ten days after childbirth. Telephone contact will be initiated within 48 to 72 hours of trial randomization and then as frequently as the dyad seems necessary. Peer volunteer have experienced fatherhood and have participated in a 12-hour training program by mentors.

Sample size estimate There is no universally accepted method for calculating sample sizes for pilot studies . However, undertaking a priori sample size calculations will enhance the utility of a pilot study. Using calculations for two independent proportions, a total pilot sample size of 28 will allow for the detection of a 15% difference in depressive symptoms scores (30% depressive symptoms rate in control group and 15% in experimental groups). However, these calculations make no allowance for attrition, why a total pilot sample size of 40 (20 per group) is recommended to allow for a 30% loss to follow-up.

The child health care nurse give information about the study to the all first time father during two months. The fathers which show interest to be included in the study will answer the EPDS. Participant inclusion criteria: Healthy baby, father aged 18 - 49 years, less than two weeks after childbirth, scored more than nine on the EPDS during last trimester in pregnancy, and Swedish or English speaking Participant exclusion criteria: current use of anti-depressant or anti-psychotic medication.

Data is collected with questionnaires. The baseline questionnaire, handed out by the child health care nurses, is completed at home and posted to the research team. A mail asking the fathers to answer a follow-up questionnaire on a study web quest will be sent out four months after the child's birth and a second follow up one year. and include follow measurement: Martial dyadic adjustment measured by Dyadic Consensus Subscale (DCS), Depressive symptoms by Edinburgh depression scale (EPDS), Anxiety measured by the The State-Anxiety Inventory (STAI), , Satisfaction with peer support, measured by study construct questions and also self-rated health.

Depressive symptoms in fathers will be measured by the Edinburgh Postnatal Depression Scale (EPDS). EPDS is a screening instrument used primarily in health care facilities to identify PPD in women . The questionnaire has been translated into several languages, including Swedish and validated on mothers and fathers. The EPDS is a 10-item four-point scale, with a total score of 0-30. A higher score indicates more depressive symptoms. All the questions in the EPDS must be answered for a person's level of depressive symptoms to be estimated. A cut-off 10 is recommended to identify the risk of post-natal depression, and a cut-off of > 11 to identify depressive illness of varying severity.

Anxiety will be measured using the Spielberger State-Anxiety Inventory (STAI-State), a 20-item self-report instrument developed to assess levels of relatively transient situation-related (state) anxiety. Items are rated on a 4-point Likert-type scale to produce a summative score ranging from 20 to 80 with higher scores indicating higher levels of anxiety. The STAI-state has been used widely in pregnancy and postpartum studies and anxiety has been consistently related to depressive symptomatology in new mothers. It is hypothesized that peer support will decrease maternal anxiety. Cronbach's alphas at 12 and weeks postpartum from pilot data were 0.94 and 0.95 respectively.

-Self reported health birth experiences and open-ended question about experiences about the program in the intervention group or parental classes in control group.

Paternal Evaluation of Peer Support will be measured using the Peer Support Evaluation Inventory, a 4- subscale self-report instrument that assesses supportive interactions, relationship qualities, perceived benefits, and satisfaction. This instrument is an enhanced version of the one used in the breastfeeding trial,89 with modifications based on Dennis' postdoctoral theoretical work. Three North American social support experts assessed content validity and preliminary psychometric testing has been completed. The Cronbach's alphas for all the subscales were above 0.91.

Peer Volunteer Evaluation of Peer Support will be assessed via telephone at the end of the trial or when a peer volunteer discontinues, will be measured using the Peer Volunteer Experience Questionnaire. Questions are related to (1) program training, (2) interactional characteristics, (3) volunteer roles, (4) personal effects, and (5) recruitment and retention.

Peer Volunteer Activities. All intervention activities (e.g., telephone discussions, left messages) will be documented by the peer volunteers using the Peer Volunteer Activity Log. The activity log was developed for the breastfeeding trial and are modified for this pilot trial. Peer volunteers will be requested to return the activity log for a supported father at 12 weeks postpartum.

Process evaluation Comprehensive process evaluation will be undertaken to explore sustainability issues and to assess intervention compliance. Intervention fidelity will be surveyed during the trial process through a questionnaire. Adherence to the study protocol will be monitored and intervention fidelity will also be secured through close contact between the research group and the mentor as soon as practical problems occurs, through telephone, email and at the follow-up workshops. The participants in the trial will also conduct evaluation of the content of the peer support since the follow-up questionnaires at four months include a number of questions about the received program. These questions will both assess fathers' experiences with the program but also ensure adherence to the study protocol.

Timelines To initiate the trial recruit fathers will take approximately three months for the pilot. Data collection for the trial is expected to take one year and the interventions will be performed during one year. Recruitment will differ between the participating clinics due to variances in size and number. After completed data collection analysis of the data according to the primary outcomes will take approximately six months. The timeline for all phases of the trial is outlined in Table 1. It is anticipated that the study will begin in September 2016 and will be completed approximately in 18 months.

Ethical concerns Since support today varies extensively between clinics and the fathers normally have no possibility of choosing model of support in the ordinary care, this should not be an ethical problem. De-identification will be made directly in connection to the collection surveys. All participants will receive a code number, this secure that individual could not identified neither during the analysis nor in the results. The information letter include Ethical approval has been sought and approved for the study by the Regional Research and Ethics Committee at Karolinska Institutet, Stockholm, 2015/1662-31.

Clinical and theoretical relevance The long-term goal of this project is to improve methods to increase the mental health among new fathers and developmental trajectories among children. The outcome of this study could provide useful clinical guidelines to identify and reduce paternal parental depressive symptoms. Instead of focusing on medical treatment by professionals, the focus will be on fathers' own capabilities. If the research team identify predictors for depressive symptoms among fathers, it could move further to develop interventions to meet fathers' needs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 49 years old,
* Less than two weeks postpartum
* Scored more than ten on the -Edingburg postnatal depression scale (EPDS ) scale <10 = indicate depression
* Swedish or English speaking

Exclusion Criteria:

- Current use of anti-depressant or anti-psychotic medication

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participant inclusion criteria on self-reported gender
Study Population: Fathers vid depressive symtoms according to EPDS more than 10 points on the scale.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-10 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Changes of Postpartum Depressive symptoms | Baseline and follow up 3 months and one year after the invention
  Changes in Postpartum Depressive symptoms (PPD), assesed by measured by EPDS (Edinburg postpartumdepression scale) more than 10 score on EPDS= indicate depressive symptoms for fathers, minimum=0 maximum=30 Postpartum Depressive symptoms (PPD), as measured by EPDS (Edinburg postnatal depression scale (Cox et al 1994)

SECONDARY OUTCOMES:
Changes of Anxiety symptoms | Baseline and follow up 3 months and one year after the invention
  Anxiety will be measured using the Spielberger State-Anxiety Inventory (STAI-State), a 20-item self-report instrument developed to assess levels of relatively transient situation-related (state) anxiety. Items are rated on a 4-point Likert-type scale to produce a summative score ranging from 20 to 80 with higher scores indicating higher levels of anxiety.

OTHER OUTCOMES:
Satisfaction with telephone peer support | follow up 3 months after the intervention
  Satisfaction with telephone peer support is assesed by measure with study construction question

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Andersson, Dr, Principal Investigator — Karolinska Institutet
Locations (1):
- Eva andersson, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No